CLINICAL TRIAL: NCT06572228
Title: AIM4: Next Step - Asthma Uncontrolled With ICS in Medium Dose (GINA 4): Next Step; Efficacy of Dupilumab Added to Medium Dose ICS/LABA in Comparison to ICS Dose Escalation to High Dose ICS/LABA in Patients With Uncontrolled Asthma
Brief Title: Efficacy of Dupilumab Added to Medium Dose Inhaled Corticosteroid/Long-acting Beta-agonist (ICS/LABA) in Comparison to ICS Dose Escalation to High Dose ICS/LABA in Adolescent and Adult Patients With Uncontrolled Asthma
Acronym: AIM4:Next Step
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R668-AS-2373; 2023-510458-18-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Asthma
Keywords: Uncontrolled; Severe exacerbations; Type 2 Inflammation; Elevated blood eosinophils; Increased Fractional exhaled Nitric Oxide (FeNO); Atopy and elevated Immunoglobulin E (IgE)
MeSH Terms: conditions — Asthma | interventions — dupilumab; Fluticasone; Propionates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dupilumab + ICS/LABA (Experimental): Randomized 1:1
  Interventions: Drug: dupilumab; Drug: ICS/LABA
- Placebo + ICS/LABA (Placebo Comparator): Randomized 1:1
  Interventions: Drug: Matching Placebo; Drug: ICS/LABA

INTERVENTIONS:
Drug: dupilumab — Administered by subcutaneous (SC) injection
  Other Names: Dupixent®; REGN668; SAR231893
  Arms: Dupilumab + ICS/LABA
Drug: Matching Placebo — Administered by SC injection
  Arms: Placebo + ICS/LABA
Drug: ICS/LABA — Administered at a blinded dose
  Other Names: fluticasone; propionate/salmeterol HFA; inhalation aerosol

SUMMARY:
This study is researching a drug called dupilumab. The study is focused on patients who have uncontrolled asthma. Asthma is a condition where the airways narrow and swell, making it difficult to breathe. Uncontrolled asthma means that patients are still having frequent symptoms while taking their current asthma medication.

The aim of the study is to see which regimen is more effective: taking dupilumab with an inhaled asthma medication or only taking a higher dose of the inhaled asthma medication. The type of asthma medication that will be used is a combination inhaled corticosteroid and long-acting beta-agonist (referred to as an ICS/LABA). Some patients may also receive an additional asthma medication called a long-acting muscarinic antagonist (referred to as a LAMA) if they are already receiving a LAMA.

The study is also looking at:

• What side effects may happen from taking dupilumab

DETAILED DESCRIPTION:
This study is a Phase 3b in Canada Minors will not be enrolled in Denmark

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of asthma for ≥12 months, based on the Global Initiative for Asthma (GINA) 2023 guidance document
2. Existing treatment with medium dose ICS/LABA (>250 to 500 μg/day of fluticasone propionate DPI or equivalent, per GINA 2023 guidance document) for at least 3 months with a stable dose ≥1 month prior to visit 1
3. Participants requiring a maximum of 3 controllers for their asthma will be considered eligible for this study
4. Pre-bronchodilator FEV1, as defined in the protocol
5. Reversibility of at least 12% and 200 mL in FEV1 after the administration of 200 to 400 μg albuterol/salbutamol at screening OR a documented history of ≥20% reduction in the FEV1, as defined in the protocol
6. Demonstrated adherence to medium dose ICS/LABA on at least 80% of days during the run-in period
7. ACQ-5 score ≥1.5 at screening (visit 1)
8. History of ≥1 severe exacerbation(s) in the previous year before visit 1, but not in the 30 days immediately preceding visit 1
9. Biomarker criteria: Baseline blood eosinophil count ≥300 cells/μL at visit 1 (~90% of population), as defined in the protocol

Key Exclusion Criteria:

1. Diagnosis of chronic obstructive pulmonary disease (COPD) or other lung diseases which may impair lung function and interfere with treatment assessments
2. Clinical evidence of lung disease(s) other than asthma or imaging (Chest X-ray, computed tomography (CT), magnetic resonance imaging [MRI]) with significant findings within 12 months of visit 1 and up to and including the baseline visit (visit 3)
3. A participant who experiences a severe asthma exacerbation at any time from 1 month prior to the screening visit (visit 1) up to and including the baseline visit (visit 3), as defined in the protocol
4. Weight is less than 30 kilograms
5. Current smoker or cessation of smoking within 6 months prior to visit 1 or previous smoker with a smoking history ≥10 pack-years
6. Severe concomitant illness(es) that, in the Investigator's judgment, would adversely affect the participant's participation in the study, as defined in the protocol
7. Participants cannot be on systemic corticosteroids at any time from 1 month prior to the screening visit (visit 1) through the duration of the run-in period

NOTE: Other protocol-defined Inclusion/Exclusion criteria apply

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Annualized severe asthma exacerbation rate | Baseline through Week 52

SECONDARY OUTCOMES:
Change in pre-bronchodilator Forced expiratory volume in the first second (FEV1) | Baseline to week 12
Annualized cumulative dose of systemic corticosteroid exposure to treat severe asthma exacerbations | Baseline to week 52
Change in Asthma Control Questionnaire (ACQ-5) | Baseline to week 12
  The ACQ-5 has 5 items that assess the most common asthma symptoms: 1. Frequency in past week awoken by asthma during the night, 2. Severity of asthma symptoms in the morning, 3. Limitation of daily activities due to asthma, 4. Shortness of breath due to asthma and 5. Wheeze. Participants are asked to recall how their asthma has been during the previous week and to respond to the symptom questions on a 7-point scale (0=no impairment, 6=maximum impairment). The ACQ-5 global score is the mean of the 5 questions and, therefore, between 0 (totally controlled) and 6 (severely uncontrolled). Higher score indicates lower asthma control.
Proportion of participants achieving ACQ-5 <1.5 | At week 12
Change in pre-bronchodilator FEV1 | Baseline up to week 52
Change in percent predicted FEV1 | Baseline up to week 52
Change in peak expiratory flow (PEF) | Baseline up to week 52
Change in forced vital capacity (FVC) | Baseline up to week 52
Change in forced expiratory flow (FEF) 25-75% | Baseline up to week 52
Change in FEV1: FVC ratio | Baseline up to week 52
Change in post-bronchodilator FEV1 | Baseline up to week 52
Time to first severe exacerbation event | Up to week 52
Proportion of participants achieving a 0.5-point improvement minimal clinically important difference (MCID) in ACQ-5 | Up to week 52
Incidence of Treatment-emergent adverse event (TEAEs) | Up to week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (84):
- United States (55):
  - Kern Research, Inc, Bakersfield, California
  - Modena Allergy & Asthma, Inc., La Jolla, California
  - Antelope Valley Clinical Trials, Lancaster, California
  - Ark Clinical Research - Long Beach, Long Beach, California
  - Newport Native Md, Inc., Newport Beach, California
  - Childrens Hospital of Orange County Main Campus, Orange, California
  - Riviera Allergy Medical Center, Redondo Beach, California
  - Raffi Tachdjian MD, Inc., Santa Monica, California
  - Bensch Clinical Research, Stockton, California
  - Integrated Research of Inland, Inc., Upland, California
  - Allianz Research Institute, Westminster, California
  - National Jewish Health, Denver, Colorado
  - St Francis Medical Institute, Clearwater, Florida
  - Florida Lung, Asthma and Sleep Specialists (FLASS) - Celebration, Kissimmee, Florida
  - Clinical Site Partners, LLC DBA Flourish Research, Winter Park, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Sneeze Wheeze and Itch Associates, Normal, Illinois
  - Asthma and Allergy Center of Chicago, River Forest, Illinois
  - NorthShore University Health System, Skokie, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Bluegrass Allergy Research, Lexington, Kentucky
  - Family Allergy and Asthma Research Institute, Louisville, Kentucky
  - Allergy & Asthma Specialists, P.S.C., Owensboro, Kentucky
  - Paul A. Shapero, M.D., Bangor, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Allergy and Asthma Center of Minnesota, Maplewood, Minnesota
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Montana Medical Research, Missoula, Montana
  - The Asthma and Allergy Center, Bellevue, Nebraska
  - Henderson Clinical Trials, Henderson, Nevada
  - Certified Research Associates, Cortland, New York
  - New York Medical College, Hawthorne, New York
  - Northwell Health at ENT & Allergy Associates, New York, New York
  - Rochester Regional Health - Alexander Park - Allergy, Immunology & Rheumatology, Rochester, New York
  - Cincinnati Childrens Hospital and Medical Center, Cincinnati, Ohio
  - Allergy Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Clinical Research Associates of Central PA, DuBois, Pennsylvania
  - University of Pittsburgh Asthma and Environmental Health Lung Institute, Pittsburgh, Pennsylvania
  - Pulmonology Associates Inc., Wynnewood, Pennsylvania
  - Dharma MD PA d/b/a Southwest Family Medicine Associates, Dallas, Texas
  - Premier Pulmonary Critical Care and Sleep Medicine, Denison, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Baylor College of Medicine - Section of Pulmonary and Critical Care, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Metroplex Pulmonary and Sleep Center, PA, McKinney, Texas
  - Lung Sleep Research Institute, North Richland Hills, Texas
  - South Texas Allergy & Asthma Medical Professionals (STAAMP) Research, San Antonio, Texas
  - Allergy & Asthma Care of Waco, Waco, Texas
  - Intermountain Medical Center - Murray (Pulmonary Medicine), Murray, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Vancouver Clinic, Vancouver, Washington
- Canada (7):
  - The Lung Centre at Vancouver General Hospital, Vancouver, British Columbia
  - Dynamic Drug Advancement Ltd., Ajax, Ontario
  - Evidence Based Medical Educator Inc., Toronto, Ontario
  - Inspiration Research Limited, Toronto, Ontario
  - Dr. Syed Anees Medicine Professional Corporation, Windsor, Ontario
  - Institut Universitare de Cardiologie et de Pneumologie de Quebec (IUCPQ) - Universite Laval, Québec
  - Clinique de Specialisee en Allergie de la Capitale, Québec
- Denmark (2):
  - Copenhagen University Hospital - Hvidovre, Hvidovre, Capital Region
  - Vejle Sygehus, Vejle, Region Syddanmark
- Germany (8):
  - Praxis fur Pneumologie am Duako, Augsburg, Bavaria
  - LMU University Hospital Munich, Munich, Bavaria
  - IKF Pneumologie Frankfurt GmbH & Co KG, Frankfurt am Main, Hesse
  - KPPK Studienzentrum, Koblenz, Rhineland-Palatinate
  - Velocity Clinical Research Lubeck GmbH (Formerly KLB Gesundheitsforschung Lübeck GmbH), Lübeck, Schleswig-Holstein
  - Lungenpraxis Hohenzollerndamm RCMS, Berlin
  - POIS Sachsen GmbH iG, Leipzig
  - IKF Pneumologie GmbH & Co. KG, Mainz
- Poland (9):
  - Centrum Medyczne All-Med, Krakow, Lesser Poland Voivodeship
  - Michał Bogacki - DOBROSTAN, Wroclaw, Lower Silesian Voivodeship
  - Diamond Clinic sp zoo, Krakow, Malopolska
  - European Trial Group (ETG) Warsaw, Warsaw, Mazovian
  - Centrum Medycyny Oddechowej Mroz SJ, Bialystok, Podlaskie Voivodeship
  - Allergy Clinic NZOZ Homeo Medicus, Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Budynek Centrum Medycyny Nieinwazyjnej, Gdansk, Pomeranian Voivodeship
  - Lekarze Specjaliści Małolepszy i Partnerzy, Wroclaw
  - ALL-MED Specjalistyczna Opieka Medyczna Medyczny Instytut Badawczy, Wroclaw
- Puerto Rico (3):
  - Allianze pulmonary Research, Guaynabo
  - Fundacion de Investigacion (FDI) Clinical Research, San Juan
  - PRCCI Clinical Research Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has :
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/